CLINICAL TRIAL: NCT04281199
Title: Multi-Institutional Pilot Study of Total Body Irradiation Using Intensity Modulated Radiation Therapy (IMRT) (VMAT or Tomotherapy) for Allogeneic HSCT With New Lung Radiation Dose Guidelines to Prevent Pul Toxicities
Brief Title: TBI Using IMRT (VMAT or Tomotherapy) for the Prevention of Pul Toxicities in Patients Undergoing Donor SCT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19508; NCI-2019-08957 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19508 (Other: City of Hope Medical Center)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Radiotherapy, Intensity-Modulated; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: Radiation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TBI, IMRT) (Experimental): Patients undergo TBI using IMRT with VMAT or tomotherapy BID on days -7 to -4 then undergo stem cell transplantation on day 0.
  Interventions: Procedure: Hematopoietic Cell Transplantation; Radiation: Intensity-Modulated Radiation Therapy; Radiation: Tomotherapy; Radiation: Total-Body Irradiation; Radiation: Volume Modulated Arc Therapy

INTERVENTIONS:
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Radiation: Tomotherapy — Undergo IMRT with tomotherapy
  Other Names: helical tomotherapy
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation
Radiation: Volume Modulated Arc Therapy — Undergo IMRT with VMAT
  Other Names: VMAT

SUMMARY:
This trial studies how well radiation therapy techniques, volumetric modulated arc therapy (VMAT) and tomotherapy, work to reduce doses to the lung compared to standard total body irradiation methods to prevent pulmonary toxicities. Standard total body irradiation is limited in its ability to spare normal organs, with only the lung being partially spared by lung blocks and risks the development of pulmonary toxicities. Reducing the doses to the lung using VMAT or tomotherapy may improve survival and decrease long term lung side effects in patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether the investigators can achieve a mean lung dose of < 8 Gy and still treat the total body at a minimum of 85% prescribed dose in patients undergoing allogeneic hematopoietic stem cell transplantation who are eligible for standard total body irradiation (TBI)-based myeloablative regimens.

II. To evaluate TBI coverage from tomotherapy and VMAT with new lung sparing guidelines.

III. To assess the rate of adverse events with intensity-modulated radiation therapy (IMRT) TBI: type, frequency, severity, attribution, time course, duration, and complications (acute graft versus host disease [GvHD], infections, and delayed neutrophil/platelet engraftment) measured by Bearman and Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

SECONDARY OBJECTIVES:

I. To evaluate dose homogeneity for all target and non-target structures using dose volume histograms.

II. To evaluate non-relapse mortality at 100 days, and 1 year post IMRT TBI. III. To evaluate relapse-free survival (RFS) at 100 days, and 1 year post IMRT TBI.

IV. To evaluate extramedullary recurrence rate at 1 year post IMRT TBI.

OUTLINE:

Patients undergo TBI using IMRT with VMAT or tomotherapy twice daily (BID) on days -7 to -4 then undergo stem cell transplantation on day 0.

After completion of study treatment, patients are followed up at 100 days and 1 year post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status (KPS) >= 70
* Acute leukemia or myelodysplastic patients evaluated within 30 days of start of conditioning regimen who would be candidates for TBI-cyclophosphamide (Cy) or TBI-etoposide (VP16) per City of Hope (COH) standard operating procedure (SOP) for allogeneic hematopoietic stem cell transplant
* Patients must be suitable for TBI conditioning regimens as part of transplant per the referring hematologist
* Patients must have adequate organ function for hematopoietic cell transplantation (HCT) as determined by the hematologist
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation
* All subjects must have the ability to understand the treatment and the willingness to sign a written informed consent
* The effects of total body radiation on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Although not mandated by the protocol, the results of the imaging scans and labs (complete blood count [CBC], comprehensive metabolic panel [CMP]) that are performed as part of the standard work up should be available and should have been done within 2 months prior to study entry
* Prior therapy (chemotherapy, immunotherapy, radiotherapy) must be completed at least 2 weeks prior to TBI
* All patients with prior radiotherapy need to be reviewed with the principal investigator (PI) to determine eligibility
* Prior therapy with chemotherapeutic agents is allowed
* DONOR: Donor evaluation and eligibility will be assessed per current COH standard operating procedure

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Prior history of radiation therapy must be presented to study PI for eligibility determination
* Pregnant women are excluded from this study because total body irradiation is an agent with the potential for teratogenic or abortifacient effects
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Completion of all fractions of intensity-modulated radiation therapy (IMRT) total body irradiation (TBI) (volume modulated arc therapy or tomotherapy) | Up to 1 year post transplant
  Will be summarized using percentage and its 95% confidence interval.

SECONDARY OUTCOMES:
Dose homogeneity for all target and non-target structures | Up to 1 year post transplant
  Will use dose volume histograms.
Rate of adverse events with IMRT TBI | Up to 1 year post transplant
  Type, frequency, severity, attribution, time course, duration, and complications will be measured by Bearman and Common Terminology Criteria for Adverse Events version 5.0. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including infection.
Rate of complications with IMRT TBI | Up to 1 year post transplant
  Will include acute graft versus host disease (aGVHD), infections, delayed neutrophil/platelet engraftment. Cumulative incidence rate will be used for aGVHD, and chronic GVHD.
Non-relapse mortality | From start of therapy until non-disease related death, or last follow-up, whichever comes first, assessed at 100 days and 1 year
  Cumulative incidence rate will be used.
Extramedullary recurrence | From start of therapy, assessed at 1 year
Relapse free survival | From start of therapy, assessed at 100 days and 1 year
  Kaplan-Meier curves will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Savita V Dandapani, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States